CLINICAL TRIAL: NCT05206643
Title: Shanghai Pudong Natural Population-based Cohort Establishment and Follow-up
Brief Title: Shanghai Pudong Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Jinqiao Community Health Service Center of Pudong new area, Shanghai (Unknown); Heqing Community Health Service Center of Pudong new area, Shanghai (Unknown); Weifang Community Health Service Center of Pudong new area, Shanghai (Unknown); Jinyang Community Health Service Center of Pudong new area, Shanghai (Unknown)
Responsible Party: Sponsor
Other Study IDs: Shanghai Pudong Cohort
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-01

CONDITIONS: Public Health
Keywords: Cohort Study; Natural Population; China

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A cohort as an area probability sample of Shanghai City

SUMMARY:
This is a community-based, prospective longitudinal epidemiologic study. Our objective is to establish a natural population-based cohort in Shanghai, China based on the latest scientific researches, preliminary findings of the project team, and a close cooperation model of the Specialist Medical Consortium.

We will focus on the information and management of health status of the general population of all ages (from birth to older age). We plan to integrate the questionnaire data and sample database information into the public health information platform, in order to establish a whole health management system across the lifespan in Chinese Natural Population.

DETAILED DESCRIPTION:
Evidence-based public health approaches to prevent various chronic diseases among population of all ages have been confirmed in recent decades. Yet barriers to implement prevention approaches persist as a result of lack of knowledge about the regularity of changes in health status of people of all ages. The purpose of this study was to learn how best to promote the adoption of evidence based public health practice related to chronic disease prevention.

The whole research plan is based on a prospective cohort study.

Our previous retrospective cohort study collected historical information of the studied cohort from 2014 to 2018 from secondary medical units, residents' community health service centers, emergency departments, and their Healthrecords. Patients' past chronic diseases such as atherosclerotic cardiovascular diseases, cancers, hypertension, diabetes, heart failure, atrial fibrillation, metabolic syndrome and other metabolic diseases, information on the history of drug use, and lifestyle (if any) were collected and sorted out. Moreover, information on various chronic disease morbidity and death among members of the cohort were also collected.

The prospective cohort building on the baseline research conducted during 2019-2020. A total of 851 parameters including physical parameters as well as genetic, biologic, demographic, and psychosocial parameters were included. Specifically, baseline research contains the following procedures:

1. Epidemiological survey: Design the Public Health and Chronic Disease Prevention and Control Questionnaire in accordance with the principles and requirements of the cohort study. On the premise of informed notification, data are collected through face-to-face interviews between the studied cohort and investigators who signed the informed consent and received uniform training. Quality control staff will review the questionnaire for quality control. The main content includes demographic sociology, lifestyle, physical exercise, daily eating habits, usage of dietary supplements, personal and family medical history, psychological assessment, and female fertility history.
2. Physical examination: the examination is performed by the clinical professional physician in the health service center. The examination content includes height, weight, blood pressure, hearing, vision, internal surgery, body fat composition (optional), chest radiography, electrocardiogram, B-ultrasound, carotid ultrasound (optional), and other imaging examinations.
3. Clinical biochemical test: fasting blood collection should be performed by all individuals upon their enrollment. The blood samples collected are tested for biochemistry, liver and kidney function, blood lipid analysis, CMV/EBV/HBV DNAs and antibodies, hsCRP, and electrolyte analysis in accordance with clinical testing requirements.
4. Biological specimen collection: collect 10ml blood samples using a health checkup, then send them to Renji sample bank for separation within 2 hours, and store in -80℃ ultra-low temperature refrigerator. The blood samples are for multi-omics and serological studies.

The follow-up would be conducted from 2020 to 2030. Through annual active (phone, face-to-face interview, etc.) and passive follow-ups, we will collect the information and management of health status of the general population of all ages. Meanwhile, we will track the various chronic diseases occurrence, death, migration, etc. in our cohort. And we will collect data that matches its baseline value, analyze the morbidity and mortality of the cohort population, and grasp the morbidity, the order of the diseases, mortality, and order of the cause of death for each disease.

ELIGIBILITY:
Inclusion Criteria:

* 0~120-year-old verified urban and rural residents in Pudong District, Shanghai
* Able to give informed consent (or has a legal designee) All the selected samples were to be interviewed.

Exclusion Criteria:

severely ill or too frail to answer; or having cognitive problems; having hearing or speaking problems; or dementia.

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Natural Chinese population
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health Status of the General Population | 10 years
  Survey on the general health of the nation in a specific time
Incidence of common chronic diseases | 10 years
  Incidence of common chronic diseases including cardio-cerebrovascular diseases, cancers and metabolic diseases were calculated by age, gender and area compared by different health management mode.
Mortality of common chronic diseases | 10 years
  Mortality of common chronic diseases including cardio-cerebrovascular diseases, cancers and metabolic diseases were calculated by age, gender and area compared by different health management mode.

SECONDARY OUTCOMES:
Normalized management rate of common chronic diseases | 10 years
  Normalized management rate of common chronic diseases
Health questionnaire | 10 years
  General health questionnaire including questions about chronic diseases, lifestyle, access to health services, comorbidities, mental health, smoke, alcohol and drugs consumption. Additional questions regarding more specific themes (ASCVD, medical aid in dying, COVID-19, etc.) will be added or adapted yearly.
  Most of the questions are individually based on previously accepted or previously used questionnaires and thus, the health questionnaire used in this project does not include a specific scale of measurement for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD,PhD, Principal Investigator — Cardiology, Ren Ji Hospital, Shanghai, China
Locations (1):
- Cardiology, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No